CLINICAL TRIAL: NCT01877096
Title: Motivational Interviewing for Colonoscopy: A Feasibility and Pilot Study
Brief Title: Motivational Interviewing for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GCO 11-1377
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal Cancer
Keywords: Motivational Interviewing; Screening Colonoscopy; Cancer Prevention
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing (Experimental): Participants will undergo a brief (20-30 minutes) motivational interviewing session after their primary care appointment
  Interventions: Behavioral: Motivational Interviewing
- Attention Control (Active Comparator): Participants will undergo a brief (20-30 minutes) attention control session after their primary care appointment
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Motivational Interviewing — A brief motivational interviewing session
  Arms: Motivational Interviewing
Behavioral: Attention Control — Participants will be asked to discuss the sources (e.g., the Internet) in which they receive information about their health. This group is designed to control for potential beneficial effects of meeting with an interventionist.
  Arms: Attention Control

SUMMARY:
The purpose of this study is to begin to examine the efficacy of a motivational interviewing intervention to increase African Americans' screening colonoscopy rates. The results from this pilot study will allow us to estimate the magnitude of the intervention and mediation effect sizes.

DETAILED DESCRIPTION:
Compared to other racial groups, African Americans have the highest colorectal cancer (CRC) morbidity and mortality rates. Screening colonoscopy can aid in the early detection and prevention of CRC. A motivational interviewing (MI) intervention holds strong promise to increase African Americans' screening colonoscopy adherence and, by doing so, decrease CRC disparities. There is a great need to conduct a randomized clinical trial (RCT) that tests the efficacy of an MI intervention to increase screening colonoscopy adherence in African Americans. The first critical and necessary step in this line of research is to pilot test such an RCT.

Objective/hypotheses: The primary objective of the proposed study is to conduct pilot testing for a future RCT which will formally test the effects of MI on screening colonoscopy adherence in African Americans. The results from this pilot study will directly inform the development of a future RCT.

Specific aims: 1) To estimate the magnitude of the MI intervention effect size; and 2) To estimate the magnitude of the mediation effect sizes (drawn from Self Determination Theory).

ELIGIBILITY:
Inclusion Criteria:

* self-identified as African American
* aged 50 years or older
* attended a non-acute visit with a primary care physician
* received a primary care physician referral for a screening colonoscopy
* deemed eligible for an open access screening colonoscopy
* agreed to have a screening colonoscopy conducted at Mount Sinai
* English speaking

Exclusion Criteria:

* Personal history of CRC or chronic GI disorder

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Screening colonoscopy completion | 6 months
  Medical chart review will be conducted 6 months after the primary care appointment in which the participants received a referral for a screening colonoscopy

SECONDARY OUTCOMES:
Psychological mediators | 5 minutes before intervention
  Psychological mediators (drawn from Self Determination Theory) Participants will complete questionnaires immediately before and after the intervention/attention control session.
Psychological mediators | 5 minutes after intervention
  Psychological mediators (drawn from Self Determination Theory) Participants will complete questionnaires immediately before and after the intervention/attention control session.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Miller, PsyD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States